CLINICAL TRIAL: NCT02951611
Title: Effects of Acupuncture Stimulation on Systemic Inflammation in Patients Undergoing Video-assisted Thoracoscopic Lobectomy Surgery
Brief Title: Effects of Acupuncture Stimulation on Systemic Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acu20161023
Record Dates: First submitted 2016-10-29; First posted 2016-11-01 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2016-10

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Sham stimulation (Sham Comparator): Put the electrodes on SI3, SJ6, PC6 and LI4 without stimulation.
  Interventions: Procedure: Sham stimulation
- Treatment: Acupuncture stimulation (Experimental): Stimulate the SI3, SJ6, PC6 and LI4 since 30 minutes before anesthesia induction until the end of operation. Stimulate again at above acupoints at 6 and 24h after operation, for 30 minutes each time. The stimulation frequency is 2/100Hz. The stimulation current is two to three times of the lowest current that the patient can feel.
  Interventions: Procedure: Acupuncture stimulation

INTERVENTIONS:
Procedure: Acupuncture stimulation — Transcutaneous electrical acupoint stimulation on SI3, SJ6, PC6 and LI4
  Arms: Treatment: Acupuncture stimulation
Procedure: Sham stimulation — Put electrodes on SI3, SJ6, PC6 and LI4 without stimulation
  Arms: Sham stimulation

SUMMARY:
60 ASA physical status I or II patients, aged 18-75 years old , scheduled for elective video-assisted thoracoscopic lobectomy surgery,will be randomized into 2 groups,with 30 patients in each group: 1. control group and 2. treatment group. Patients in treatment group will receive transcutaneous electrical acupoint stimulation(TEAS) during the surgery and at 6h and 24h after surgery. Patients in the control group received only TIVA general anesthesia and sham electrical stimulation. Serum from patients of both groups will be collected at before surgery, 1h and 25h after surgery, respectively. Serum levels of TNF-alpha, IL-1 beta, CXCL8, IFN gamma and IL-4 at different time points will be measured and compared between the two groups.

DETAILED DESCRIPTION:
60 ASA physical status I or II patients, aged 18-75 years old , scheduled for elective video-assisted thoracoscopic lobectomy surgery,will be randomized into 2 groups,with 30 patients in each group: 1. control group, who will receive total intravenous anesthesia(TIVA) and sham stimulation; and 2. treatment group, who will receive (TIVA) and transcutaneous electrical acupoint stimulation(TEAS). Since 30 min before induction of anesthesia, patients in treatment group will be stimulated at the 4 acupoints , Houxi、Zhigou、Neiguan and Hegu on both sides by Han's Acupoint Nerve Stimulator(HANS) until the end of the operation. At 6h and 24h after surgery, patients in treatment group will receive TEAS again, for 30 min each time.The frequency was 2/100Hz,the stimulate intensity was the maximum current that could be tolerated when the patients were awake.The control group received only TIVA general anesthesia and sham electrical stimulation.Serum from patients of both groups will be collected at before surgery, 1h and 25h after surgery, respectively and serum levels of TNF-alpha, IL-1 beta, CXCL8, IFN gamma and IL-4 at different time points will be measured. The primary outcome measures are serum TNF-alpha and IL-1 beta levels at 25h after surgery. The secondary outcome measures include serum levels of TNF-alpha, IL-1 beta, CXCL8, Th1/Th2 ratio (by calculating IFN gamma/IL-4) at 1h post surgery and serum levels of CXCL8, Th1/Th2 ratio at 25h post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed Non-Small Cell Lung Carcinoma (NSCLC) and will have elective video-assisted thoracoscopic lobectomy surgery
* ASA grade 1-2
* BMI between 18 to 31 kg/m2

Exclusion Criteria:

* with a history of thoracic surgery
* Unwilling to receive transcutaneous electrical acupoint stimulation
* BMI ≥ 32 kg/m2
* Infection or scars at the acupoints
* periphery nerve injury at the upper or lower limbs
* Severe liver, renal, brain or lung disease
* Drug abuse
* Patients who cannot coordinate with investigators, such as dysphasia，severe infectious disease and disturbance of consciousness
* Patients participating other trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
serum TNF-α level | at 25 hour after surgery
serum IL-1β level | at 25 hour after surgery

SECONDARY OUTCOMES:
serum TNF-α level | at 1 hour after surgery
serum IL-1β level | at 1 hour after surgery
serum CXCL8 level | at 1 hour after surgery
serum CXCL8 level | at 25 hour after surgery
serum Th1/Th2 ratio | at 1 hour after surgery
serum Th1/Th2 ratio | at 25 hour after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided